CLINICAL TRIAL: NCT02473484
Title: Search of Protein Biomarkers in Order to Achieve a Molecular Classification of Gliomas
Acronym: GLIOMIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_27; 2014-A00185-42 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Glioblastoma
Keywords: High Grade Glioma; Proteomics; MALDI-MSI
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumoral DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim is to classify high grade glioma by matrix-assisted laser desorption/ionization mass spectrometry imaging (MALDI MSI). In order to provide more specific informations for the diagnosis and the prognosis of high grade glioma.

ELIGIBILITY:
Main inclusion criteria:

* Patients with grade III or IV glioma newly diagnosed with histological evidence
* Surgical indication
* Tumor tissue available at biobank of Lille
* Men and women aged ≥ 18 years
* Informed Consent signed by the patient or his legal representative.

Main exclusion criteria:

* Antecedents of other cancers except basal cell skin cancer or carcinoma in situ of the uterus cervix
* Previous history of brain radiotherapy
* Anti-tumor systemic treatments (chemotherapy or targeted therapy) prior to surgery of glioma
* Genetic disease that may cause brain tumor, potentially radiation-induced tumor
* History of degenerative neurological disease prior to diagnosis
* contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: high grade glioma
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2014-06-24 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the correlation between the WHO classification 2007 only established standard diagnostic and classification by mass spectrometry gliomas (lipids, peptides, proteins) | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Le RHUN, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Le Rhun, Lille, France

IPD SHARING:
Plan to Share IPD: No